CLINICAL TRIAL: NCT01493323
Title: Neuro Anatomic Basis of Psychic Pain in Depression and Suicidal Behaviour
Brief Title: Functional Imaging of Psychic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult to patient inclusion
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Geneva (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UF 8555
Record Dates: First submitted 2011-11-10; First posted 2011-12-15 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Suicide, Attempted; Mood Disorder
Keywords: Psychic pain; Social exclusion; Mood disorders; Suicide, attempted; Magnetic Resonance Imaging, Functional; Genetic; Physic pain
MeSH Terms: conditions — Suicide, Attempted; Mood Disorders; Social Isolation | interventions — mycophenolic adenine dinucleotide; PALM protein, human; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Experimental)
  Interventions: Behavioral: Assessment of personality traits; Behavioral: Assessment of suicidal act; Behavioral: Assessment of depression; Procedure: Cyber ball game; Procedure: Iowa Gambling Task; Procedure: Microcomputer; Procedure: blood sample
- Depressive attempters (Experimental)
  Interventions: Behavioral: Assessment of personality traits; Behavioral: Assessment of suicidal act; Behavioral: Assessment of depression; Procedure: Cyber ball game; Procedure: Iowa Gambling Task; Procedure: Microcomputer; Procedure: blood sample

INTERVENTIONS:
Behavioral: Assessment of personality traits — suicide behaviour , psychic pain, social exclusion, decision making...
  Other Names: impulsivity; anger; anxiety; emotional lability; self-administered questionnaires
Behavioral: Assessment of suicidal act — suicide behaviour , psychic pain, social exclusion, decision making...
  Other Names: SIS; RRRS
Behavioral: Assessment of depression — suicide behaviour , psychic pain, social exclusion, decision making...
  Other Names: BDI; HAMD-21
Procedure: Cyber ball game — functional neuroimaging
  Other Names: fIRM
Procedure: Iowa Gambling Task — functional neuroimaging
Procedure: Microcomputer — functional neuroimaging
  Other Names: palm
Procedure: blood sample — blood sample

SUMMARY:
Suicidal behaviour (SB) represents a major public health problem, costing life in more that one million people every year worldwide. Even if SB is considered as a consequence of social adversity and depression, these stress factors are often necessary but not sufficient to explain the occurrence of a suicidal act. A preliminary study suggests that an increased perception of psychic pain during a major depressive disorder increases the risk of suicide behaviour. The investigators aimed to investigate the relationship between social exclusion (a classic trigger of psychic pain) and SB and improve our knowledge about the physiopathology of this domain.

DETAILED DESCRIPTION:
Suicide behaviour (SB) represents a major public health problem. In order to improve prevention strategies, a better understanding of the physiopathology of SB is needed. According to a "stress vulnerability" model, people who make a suicide attempt when they are subject to a stress factor (environmental stress, interpersonal difficulties, depression, tobacco, substance abuse...) are those who have a specific vulnerability. Vulnerability factors to SB may be considered in clinical terms (propensity to hopelessness, aggressive impulsivity traits), neurobiological terms (serotoninergic system disorder, especially in the ventral prefrontal cortex-vPFC) and cognitive terms (decision making, cognitive functions mediated by the vPFC and the serotoninergic system). Finally, genetic factors seem also involved in suicide vulnerability. The investigators have conducted a preliminary study which suggests that increased perception of psychic pain during a major depressive disorder increases suicidal ideation and suicidal act. Study about anatomic basis of psychic pain and its triggers represents a relevant theme to understand the suicidal process. Among the classical factors triggering psychic pain and suicidal act, events of social exclusion appears to be crucial. Finally, many data suggests the close relationship between physic and psychic pain.

ELIGIBILITY:
Non specific criteria, for all the participants:

* Woman- 18-50 years old
* Non menopausal
* Right-handed
* Caucasian from western Europe (exception of Basque and Sardinian), for genetic purposes
* Subject who signed informed consent
* Able to understand the nature, the aim, and the methodology of the study and agree to cooperate during clinical and radiological evaluation

Specific criteria:For depressed suicide attempters :

* DSM IV criteria for major depressive disorder
* Personal history of suicide attempt
* No psychotropic treatment currently

For depressed affective controls :

* DSM IV criteria for major depressive disorder
* No personal history of suicide attempt
* No psychotropic treatment currently

For non depressed suicide attempters :

* Personal history of unipolar or bipolar mood disorder, according to DSM IV criteria
* Normothymic currently (HAMD<7)
* Personal history of suicide attempt
* Minimum treatment Healthy controls :
* No personal history of axis I psychiatric disorders according to the MINI and the DSM IV criteria

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cerebral regions associated with psychic pain during a major depressive disorder | One day
  Magnetic Resonance Imaging to visualize cerebral regions associated with psychic pain during a major depressive disorder
Cerebral regions associated with perception of social exclusion | One day
  Magnetic Resonance Imaging to visualize the cerebral regions associated with perception of social exclusion

CONTACTS AND LOCATIONS:
Overall Officials: Philippe PC Courtet, Professor(MD-PhD), Principal Investigator — University Hospital, Montpellier
Locations (1):
- MontpellierUniversity Hopital, Montpellier, France